CLINICAL TRIAL: NCT04857697
Title: Engineering Gut Microbiome to Target Cancer-Immune Microenvironment in Breast and Lung Cancer
Brief Title: Effects of Probiotics on the Gut Microbiome and Immune System in Operable Stage I-III Breast or Lung Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC210302; NCI-2021-03139 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20-011177 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Adenocarcinoma; Stage I Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Biopsy; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Supportive care (biospecimen collection, probiotic) (Experimental): Patients undergo collection of blood samples at baseline and time of surgery, and collection of stool samples at baseline and after completion of probiotic regimen. Patients receive probiotics PO once on day 1, and then BID or TID for 2-4 weeks before standard of care surgery. Patients also undergo collection of tissue samples during standard of care surgery.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Probiotic; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood, stool, and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected
Drug: Probiotic — Given PO
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery

SUMMARY:
This clinical trial evaluates whether engineering gut microbiome using probiotics will alter the body's immune system to react to stage I-III breast or lung cancers that can be removed by surgery (operable). Having diverse species of bacteria inside the bowel may help improve the immune system, particularly the ability of the immune system to recognize cancer. Taking probiotics may change the diversity and make up of the bacteria in the bowels, and change how the immune system reacts to breast or lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a pilot study of probiotics prior to surgery in operable breast and lung cancer patients.

II. To evaluate systemic and intratumoral immunomodulatory effects of probiotics in operable breast and lung cancer patients.

OUTLINE:

Patients undergo collection of blood samples at baseline and time of surgery, and collection of stool samples at baseline and after completion of probiotic regimen. Patients receive probiotics orally (PO) once on day 1, and then twice daily (BID) or three times daily (TID) for 2-4 weeks before standard of care surgery. Patients also undergo collection of tissue samples during standard of care surgery.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Histologically confirmed adenocarcinoma of the breast operable stage I-III or histologically confirmed carcinoma of the lung operable stage I-III will be enrolled prior to their definitive surgery
* Patients must have adequate organ function
* Patients must be willing to provide tissue, blood and stool samples for the research study

Exclusion Criteria:

* Patients must not receive systemic neoadjuvant therapy
* Patients must not have taken any probiotics in the past 30 days prior to the enrollment
* Patients with autoimmune disease, immune deficiency such as human immunodeficiency virus (HIV), irritable bowel, known diverticulosis, and other serious gastrointestinal (GI) conditions at treating physician's discretion will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Length and adherence of probiotics | Up to 4 weeks
  Will be collected via study diaries.
Percentage of CD8+, CD4+, and T-reg cells | Baseline up to 4 weeks
Cytokine counts | Baseline up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Saranya Chumsri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States